CLINICAL TRIAL: NCT03407404
Title: Ketamine-Midazolam Versus Morphine-Midazolam for Continous Patient Sedation in Intensive Care Units in Uganda. A Randomised Controlled Trial.
Brief Title: Comparing Clinical Outcomes Between Ketamine-midazolam and Morphine-midazolam for Continous Sedation in ICU Patients.
Acronym: KeMiMof
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Makerere University (Other)
Collaborators: THRiVE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/HD07/1275U
Record Dates: First submitted 2017-06-05; First posted 2018-01-23 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either receive ketamine-midazolam or morphine-midazolam for continous sedation at enrollment, then followed up for outcomes.
Who Masked: Participant, Investigator
Masking Description: Drugs will be premixed and coded for ketamine-midazolam or morphine-midazolam. The colorless drug mixture shall be provided to the attending physician to start the infusion at 2ml/hour and to be titrated to the desired level of sedation.
  The investigator and participant will be unaware of which group a certain patient is under.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine-midazolam (Experimental): Continous intravenous sedation with a colorless drug mixture in 50ml syringe containing 900mg ketamine and 36mg midazolam.
  Interventions: Combination Product: Ketamine-Midazolam
- Morphine-Midazolam (Active Comparator): Continous intravenous sedation with a colourless drug mixture in 50ml syringes containing 54mg morphine and 36mg midazolam.
  Interventions: Combination Product: Morphine -Midazolam

INTERVENTIONS:
Combination Product: Ketamine-Midazolam — Continous intravenous sedation with 36mg of Midazolam and 900mg of Ketamine mixed in 50ml syringes as long as patient still requires sedation.
  Arms: Ketamine-midazolam
Combination Product: Morphine -Midazolam — Continous intravenous sedation with 54mg of Morphine Sulphate and 36mg of midazolam mixed in 50ml syringes as long as participant still requires sedation.
  Arms: Morphine-Midazolam

SUMMARY:
A prospective, double-blinded, multicenter randomized control trial. All critically ill patients above 12 years of age requiring continuous sedation for >24hrs in the ICU will be screened and those meeting selection criteria (and consented) will be enrolled into the study.

.

DETAILED DESCRIPTION:
165 participants shall be consecutively randomized into either sedation with ketamine-midazolam or morphine-midazolam group using a block sequence technique; group concealed in brown envelopes. Blinding will be at patient/next of kin level as well as investigator/data collector level.

Enrolled subjects shall be followed up for treatment history, co-morbidities and related data will be collected, results analyzed and study findings will be availed to ICU physicians and Ministry of health to guide treatment considerations and for health care planning.

Data shall be collected using a standardized questionnaire by trained research assistants. It will be double entered into Epidata and exported to STATA version 12.0 for analysis. Continuous variables will be expressed as means and standard deviations, while categorical data will be expressed as frequencies with their respective percentages. Linear regression and logistic regression used to analyse primary outcomes, as well as multivariate analysis to detect associations.

ELIGIBILITY:
Inclusion Criteria:

1. Age >12years of age.
2. Anticipated need for sedation for >24hours.

Exclusion Criteria:

1. Hypertensive crisis i.e. sustained SBP >200mmHg/DBP>110mmHg
2. Status epilepticus
3. Ischemic heart disease and severe LV dysfunction
4. Persistent tachyarrythmias
5. History of mental illness
6. Hypersensitivity to ketamine, morphine or midazolam.
7. Tetanus -due to the muscle rigidity that may be caused by ketamine. Reasons for exclusions 1 to 4; Ketamine stimulates the sympathetic nervous system causing transient increase in myocardial work and blood pressure and has psychoactive effects

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation | 14 days
  in hours from start of mechanical ventialtion
incidence of hypotension | 14 days
  incidence of hypotension requiring vasopressor support.
incidence of delirium | 14 days
  assessed daily with the CAM-ICU score

SECONDARY OUTCOMES:
ICU length of stay | 14 days
  length of stay in the intensive care unit from enrollment.
mortality rate | within 14 days
  number of deaths in each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Christine Namata, MBChB, Principal Investigator — Makerere University
Locations (1):
- Mulago National Referral Hospital ICU, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No